CLINICAL TRIAL: NCT00274911
Title: Hyperfractionated Accelerated Radiotherapy (HART) With Chemotherapy (Cisplatin, CCNU, Vincristine) for Non-Pineal Supratentorial Primitive Neuroectodermal Tumours
Brief Title: Radiation Therapy Followed By Combination Chemotherapy in Treating Young Patients With Supratentorial Primitive Neuroectodermal Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-CNS-2004-01; CDR0000454540 (Registry Identifier: PDQ (Physician Data Query)); EU-20580
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood supratentorial primitive neuroectodermal tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Cisplatin; Lomustine; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: lomustine
Drug: vincristine sulfate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as lomustine, cisplatin, and vincristine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy followed by combination chemotherapy after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving radiation therapy followed by combination chemotherapy works in treating young patients with supratentorial primitive neuroectodermal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of hyperfractionated accelerated radiotherapy (HART) in pediatric patients with nonpineal supratentorial primitive neuroectodermal tumors.

Secondary

* Determine overall and relapse-free survival of patients treated with HART followed by adjuvant combination chemotherapy comprising lomustine, cisplatin, and vincristine.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Radiotherapy: Patients undergo hyperfractionated accelerated radiotherapy (HART) twice a day, 5 days a week, for 5 weeks.
* Adjuvant combination chemotherapy: Six weeks after the last radiotherapy dose, patients receive oral lomustine once and cisplatin IV over 6 hours on day 1 and vincristine IV on days 1, 8, and 15 . Treatment repeats every 6 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven nonpineal supratentorial primitive neuroectodermal tumors

  * No supratentorial atypical teratoid/rhabdoid tumors or medulloepitheliomas
* Localized or metastatic disease

  * Metastatic disease is defined as unequivocal evidence of supratentorial metastases and/or spinal metastases on pre-operative or postoperative MRI scan OR tumor cells seen on cytospin analysis of lumbar cerebrospinal fluid (stage M1) performed between 15 days and 21 days after surgery
* Has undergone surgical resection within the past 4-6 weeks

PATIENT CHARACTERISTICS:

* Able to cooperate with twice daily fractions of radiotherapy
* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Neurologically stable (or improving) during the week before starting radiotherapy
* Lansky performance status 30-100% (for patients 1 to 16 years of age) OR
* Karnofsky performance status 30-100% (for patients over 16 years of age)
* Must be able to comply with the chemotherapy protocol (e.g., no hearing loss, renal impairment)
* No presence of active uncontrolled infection
* No previous malignant disease
* Not pregnant or nursing
* No syndrome with recognized potential for increased sensitivity to radiotherapy and/or chromosomal fragility

PRIOR CONCURRENT THERAPY:

* No previous chemotherapy or radiotherapy
* The patient should not be receiving steroids, if possible, at the start of radiotherapy or should be on a stable or reducing dose of steroids during the week before starting radiotherapy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-02; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity measured by hematological, gastrointestinal, mucosal, neurological, and skin morbidity during treatment and for 6 weeks after completion of treatment

SECONDARY OUTCOMES:
Overall and relapse free survival at follow up every 2 months for 1 year, every 3 months for 2 years, and then every 6 months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank Saran, MD, Study Chair — Royal Marsden NHS Foundation Trust; Christopher Chandler, MD — King's College Hospital NHS Trust; Roger Taylor, MD — Cookridge Hospital; David Ellison, MD — Northern Centre for Cancer Treatment at Newcastle General Hospital; Barry Pizer, MD — Royal Liverpool Children's Hospital, Alder Hey
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales